CLINICAL TRIAL: NCT01064466
Title: Explore the Relationship Between Single Nucleotide Polymorphisms and Etoposide Response and Toxicity in Patients With Small Cell Lung Cancer.
Brief Title: Pharmacogenomics ANDA SNP Clinical Study - Etoposide and Single Nucleotide Polymorphisms
Acronym: Drugs-SNPs
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., Sponsor-Investigator, Medical Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IND 178172 Commercial; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); NPI - 1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI - 1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); IND 178172 (Registry Identifier: FDA IND)
Record Dates: First submitted 2010-02-02; First posted 2010-02-08 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; Etoposide; SNP; Topo; CYP; Genotype; Oncology; Genetics; Lung; Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: * The usual approach group (Oral)
  * The study approach group (Oral) (China Import)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ETOPOSIDE - Usual (Experimental): * Etoposide Capsule
  * Chemotherapy
  * Etoposide Capsule
  * Usual Approach Group
  Interventions: Drug: ETOPOSIDE - Usual
- ETOPOSIDE - Study (Experimental): * China Import Etoposide Capsule
  * Chemotherapy
  * China Import Etoposide Capsule
  * Study Approach Group
  Interventions: Drug: ETOPOSIDE - Study

INTERVENTIONS:
Drug: ETOPOSIDE - Usual — Etoposide Capsule
  Other Names: Usual Etoposide Capsule Chemotherapy
  Arms: ETOPOSIDE - Usual
Drug: ETOPOSIDE - Study — China Import Etoposide Capsule
  Other Names: Study Etoposide Capsule Chemotherapy
  Arms: ETOPOSIDE - Study

SUMMARY:
Explore the relationship between drug target topoisomerase II gene single nucleotide polymorphisms and Etoposide (VP-16) therapeutic-effects in patients with small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

Explore the relationship between drug target CYP4503A4 gene single nucleotide polymorphisms and Etoposide (VP-16) side-effects in patients with small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

DETAILED DESCRIPTION:
The usual approach group, after lung tissue biopsy, 300 double blind random group separated SCLC patients currently used the Chemotherapy on ETOPOSIDE capsule, it will try to look for the relationship between the ETOPOSIDE therapeutic efficacy and the Topoisomerase II SNP Genotyping, and the relationship between the ETOPOSIDE therapeutic safety and the CYP4503A4 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

The study approach group, after lung tissue biopsy, 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Etoposide Capsule, it will try to look for the relationship between the ETOPOSIDE therapeutic efficacy and the Topoisomerase II SNP Genotyping, and the relationship between the ETOPOSIDE therapeutic safety and the CYP4503A4 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

* 1) Detect drug target whole gene precision sequence of everyone patient for all 600 recruited double blind SCLC patients.
* 2) Mutually compare everyone patient drug target whole gene precision sequence for a total of 600 recruited double blind SCLC patients.
* 3) Calculate drug target gene SNPs in all 600 recruited double blind SCLC patients.
* 4) Correlate everyone patient drug target gene SNP to everyone patient drug efficacy.
* 5) Correlate everyone patient drug target gene SNP to everyone patient drug safety.
* 6) Mutually compare the usual approach group SNPs (300 double blind random group separated SCLC patients) with the study approach group SNPs (300 double blind random group separated SCLC patients).
* 7) Confirm the relationship between drug target gene SNPs and drug efficacy.
* 8) Confirm the relationship between drug target gene SNPs and drug safety.

ELIGIBILITY:
* Select 600 Small Cell Lung Cancer Patients who are suitable for lung tissue biopsy
* Dosage Duration at least 45 days
* The usual approach group - Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on Etoposide Capsule after lung tissue biopsy, like as the usual approach group.
* The study approach group - Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Etoposide Capsule after lung tissue biopsy, like as the study approach group.

The inclusion criteria:

* 1. Clinical diagnosis of Small Cell Lung Cancer (SCLC)
* 2. Clinical lung tissue biopsy diagnosis of SCLC
* 3. Suitable for enough lung tissue biopsy of SCLC
* 4. Random and double blind
* 5. Measurable disease
* 6. Adequate organ functions
* 7. Adequate performance status
* 8. Age 24 years old and over
* 9. Sign an informed consent form
* 10. Receive blood-drawing

The exclusion criteria:

* 1. Pneumonectomy
* 2. Treatment with other anti-cancer therapies and cannot be stopped currently
* 3. Pregnancy
* 4. Breast-feeding
* 5. The patients with other serious intercurrent illness or infectious diseases
* 6. Have more than one different kind of cancer at the same time
* 7. Serious Allergy to Drugs
* 8. Clot or Bleed Tendency
* 9. Serious Risks or Serious Adverse Events of the drug product
* 10. The prohibition of drug products
* 11. Have no therapeutic effects
* 12. Follow up to the most current label

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Find Etoposide Drug Targets' SNP Genotypes which are effectiveness-associated, and which are risk-associated. | Duration at least 90 days
  1. Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on Etoposide Capsule after lung tissue biopsy, like as the usual approach group.
  2. Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Etoposide Capsule after lung tissue biopsy, like as the study approach group.
  3. Assay above every SCLC patient-specific Etoposide (VP-16) drug target (Topoisomerase II) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  4. Assay above every SCLC patient-specific Etoposide (VP-16) drug target (CYP4503A4) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. (MIDI) - IORG0007849 - NPI 1023387701; HAN XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. (MIDI) - IORG0007849 - NPI 1023387701; HAN XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. (MIDI) - IORG0007849 - NPI 1023387701
Locations (1):
- Medicine Invention Design, Inc. (MIDI) - IORG0007849 - NPI 1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWA < 00015357 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IRB < 00009424 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IORG < 0007849 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT01064466/Prot_019.pdf
  • Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT01064466/SAP_020.pdf
  • Informed Consent Form (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT01064466/ICF_021.pdf